CLINICAL TRIAL: NCT03943264
Title: Phase 1b Open-Label, Dose-Identification Study of XPro1595 in Patients With Alzheimer's Disease and Biomarkers of Inflammation.
Brief Title: A Biomarker-directed Study of XPro1595 in Patients With Alzheimer's
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inmune Bio, Inc. (Industry)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XPRO1595-AD; 18PTC-R-592167 (Other Grant/Funding Number: Alzheimer's Association)
Record Dates: First submitted 2019-04-26; First posted 2019-05-09 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Alzheimer Disease
Keywords: inflammation; Biomarker; TNF
MeSH Terms: conditions — Alzheimer Disease; Inflammation | interventions — XENP 1595

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.3 mg/kg XPro1595 (Experimental): 0.3 mg/kg of XPro1595 will be administered via subcutaneous injection once a week for 12 weeks.
  Interventions: Drug: XPro1595
- 0.6 mg/kg XPro1595 (Experimental): 0.6 mg/kg of XPro1595 will be administered via subcutaneous injection once a week for 12 weeks.
  Interventions: Drug: XPro1595
- 1.0 mg/kg XPro1595 (Experimental): 1.0 mg/kg of XPro1595 will be administered via subcutaneous injection once a week for 12 weeks.
  Interventions: Drug: XPro1595

INTERVENTIONS:
Drug: XPro1595 — XPro1595 will be delivered by subcutaneous injection once a week
  Other Names: INB03, DN-TNF, XENP345

SUMMARY:
The purpose of this study is to evaluate safety and target engagement of XPro1595 in Alzheimer's patients with biomarkers of inflammation.

DETAILED DESCRIPTION:
The study is designed as a multicentre, phase 1b open-label study. The objectives of this study are to determine the safety, tolerability, and efficacy of XPro1595 in patients with Alzheimer's disease and at least one of the following inflammatory biomarkers: high sensitivity c-reactive protein (hs-CRP), hemoglobin A1c, erythrocyte sedimentation rate (ESR), or one Apolipoprotein E4 allele.

XPro1595 is a second-generation inhibitor of tumor necrosis factor (TNF) that selectively neutralizes soluble TNF, an inflammatory factor implicated in Alzheimer's pathology.

A key element of this study is to identify Alzheimer's patients that are most likely to benefit from XPro1595 treatment. Enrollment is limited to patients with evidence of inflammation. For instance, hs-CRP is an inflammatory biomarker elevated in the blood of some Alzheimer's patients and elevated CRP has been shown to predict response to TNF inhibitors in multiple other diseases.

Alzheimer's patients with elevated inflammatory biomarkers will be enrolled in a 12-week study to determine the safety and the ability of XPro1595 to reduce neuroinflammation using a combination of invasive and non-invasive biomarkers of inflammation. The study will identify the dose of XPro1595 to be used in a larger Phase II disease modification study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and above at screening;
2. Diagnosed with probable AD defined by the National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association criteria;
3. Has hsCRP levels ≥1.5mg/L,OR HbA1c ≥ 6DCCT %, OR Erythrocyte Sedimentation Rate (ESR) ≥10 mm/h, OR APOE4 positive (at least one APOE4 allele);
4. Female of childbearing potential (FCBP) must have confirmed negative urine pregnancy test at Screening;
5. All female of childbearing potential (FCBP) and male patients who are sexually active with a female of childbearing potential must agree to use a highly effective contraception during the treatment period and until 90 days after the last dose of treatment for sexually active males whose partners are FCBP or until 30 days after the last dose of treatment for FCBP.
6. Consents to having lumbar punctures;
7. Consents to apolipoprotein E (APOE) genotyping(if status unknown);
8. Provide written informed consent prior to any study procedures being performed;
9. Has a caregiver who either lives in the same household or interacts withthe patient at least 4 hours per day and at least 4 days per week, who is knowledgeable about the participant's daytime and night-time behaviours and who canbe available to attend all clinic visits in personat which caregiver assessments are performed.Patients with caregivers that do not meet this criterionbut are determined by the investigator as able to provide an adequate assessment of the patient may also participate with prior approval from the sponsor.

Exclusion Criteria:

1. Patients taking cholinesterase inhibitors, memantine, or antidepressant medication for less than 45 days from Day 1 (i.e. must be on stable dose for at least 45 days prior to Day 1);
2. Have taken within the last 45 days from Day 1; corticosteroids or other immunosuppressive drugs, thalidomide or other TNF active drugs, minocycline.
3. Enrolled in another clinical trial where patients receive treatment with investigational drug or device or have received treatment on another AD clinical trial within the last 60 days from Day 1;
4. Unable to tolerate lumbar puncture or taking medicine where lumber punctures are contraindicated (anti-coagulants besides daily 100mg of aspirin);
5. A prior organ or stem cell transplant;
6. A major adverse cardiac event within 6 months before screening;
7. Lymphoma, leukaemia, or any malignancy within the past 5 years with the exception of malignancies with negligible risk of metastasis or death, such as basal cell or squamous cell carcinomas of the skin or cervical carcinoma in situ that have been resected with no evidence of metastatic disease for 3 years;
8. Jaundice, active hepatitis, or known hepatobiliary disease (except asymptomatic cholelithiasis);
9. Positive screening assessment for viral hepatitis B surface antigen or hepatitis C virus (HCV) antibody and positive HCV ribonucleic acid or human immunodeficiency virus, or a history of illicit drug injecting;
10. Seated blood pressure of ≥ 165/105 mmHg at screening;
11. Unable to comply with the study procedures and assessments;12.Known hypersensitivity to investigational product or its excipients;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
The number of patients with a treatment-emergent adverse event throughout 12 weeks of treatment with XPro1595 | 12 weeks
  Adverse events will be assessed by clinical and laboratory measures
The percentage of patients with a treatment-emergent adverse event throughout 12 weeks of treatment with XPro1595 | 12 weeks
  Adverse events will be assessed by clinical and laboratory measures

SECONDARY OUTCOMES:
Changes from baseline in high sensitivity C-reactive protein in the blood and cerebral spinal fluid following 12 weeks of treatment with XPro1595 | 12 weeks
  To compare changes in high sensitivity C-reactive protein
Changes from baseline in inflammatory cytokines in the blood and cerebral following 12 weeks of treatment with XPro1595 spinal fluid | 12 weeks
  To compare changes in Inflammatory cytokines; including but not limited to tumor necrosis factor, interleukin-1, and interleukin-6
Changes from baseline in blood and cerebral spinal fluid levels of amyloid beta following 12 weeks of treatment with XPro1595 | 12 weeks
  To compare changes in amyloid in cerebral spinal fluid
Changes from baseline in cerebral spinal fluid levels of tau following 12 weeks of treatment with XPro1595 | 12 weeks
  To compare changes in tau in cerebral spinal fluid
Change from baseline in FreeWater content (edema) using magnetic resonance imaging following 12 weeks of treatment with XPro1595 | 12 weeks
  To compare changes in FreeWater content as a proxy of neuroinflammation following 12 weeks of treatment with XPro1595
Change from baseline in the Mini-Mental State Examination (MMSE) following 12 weeks of treatment with XPro1595 | 12 weeks
  The Mini-Mental State Examination (MMSE) provides a comprehensive measure of cognitive function. The maximum possible score is 30 and patients scoring below 23 are classified as having cognitive impairment as follows, mild (19 to 23), moderate (10 to 18), severe (below 9).
Change from baseline in the Digit Symbol Substitution Test (DSST) following 12 weeks of treatment with XPro1595 | 12 weeks
  The Digit Symbol Substitution Test (DSST) is a cognitive test that consists of digit-symbol pairs. The patient records the corresponding symbol to each presented digit in 90 seconds. The total number of correct symbols is counted to provide a score between 0 and 133. Higher scores indicate better cognitive functioning.
Change from baseline in the Verbal Fluency Test following 12 weeks of treatment with XPro1595 | 12 weeks
  In the Verbal Fluency Test, patients are given a letter and asked to name as many words as they can that begin with that letter in 60 seconds. The number of correct responses is counted. A higher number of responses indicates better cognitive functioning.
Change from baseline in the Neuropsychiatric Inventory (NPI) following 12 weeks of treatment with XPro1595 | 12 weeks
  Neuropsychiatric Inventory (NPI) is a measure of frequency and severity of common psychiatric symptoms related to dementia using a 12-question measure. For each question, a score is given for frequency, severity and caregiver distress. Total scores range from 0 to 144. A higher score means greater neuropsychiatric disturbance.
Change from baseline in the Bristol Activities of Daily Living Scale (BALDS) following 12 weeks of treatment with XPro1595 | 12 weeks
  Bristol Activities of Daily Living Scale (BADLS) is a questionnaire that measures the impact of Alzheimer's disease on daily activities using a 20-item questionnaire. Total scores range from 0 to 60. A higher score indicates a greater disturbance in daily living.
Change from baseline in the Memory-Enhanced Retrospective Evaluation of Treatment Observer Reported Global Impression of Improvement (MERET OBSRO-C) following 12 weeks of treatment with XPro1595 | 12 weeks
  Memory-Enhanced Retrospective Evaluation of Treatment Observer Reported Global Impression of Improvement (MERET OBSRO-C) evaluates caregivers' self-reports of treatment efficacy with self-prompted memory aids regarding their clinical experiences obtained prior to treatment initiation.
Evaluate changes in the Memory-Enhanced Retrospective Evaluation of Change from baseline Global Impression of Improvement (MERET PGI-C) following 12 weeks of treatment with XPro1595 | 12 weeks
  Memory-Enhanced Retrospective Evaluation of Treatment Patient Global Impression of Improvement (MERET PGI-C) evaluates patients self-reports of treatment efficacy with self-prompted memory aids regarding their clinical experience obtained prior to treatment initiation. Patient's global impression of (PGI-I) ratings will be obtained using a web-based interface prior to and following playback of impromptu patient recordings obtained prior to the start of treatment (MERET).

OTHER OUTCOMES:
Change from baseline in Breath volatile organic compounds (BVOCs) following 12 weeks of treatment with XPro1595 | 12 weeks
  Breath volatile organic compounds (BVOCs) is a non-invasive method of measuring biological processes in exhaled breath that can be used to inform on disease and treatment-related states.

CONTACTS AND LOCATIONS:
Overall Officials: Terrence O'Brien, MD, Principal Investigator — The Alfred
Locations (5):
- Australia (5):
  - KaRa MINDS, Macquarie Park, New South Wales
  - Mater Medical Research Institute, Brisbane, Queensland
  - Central Adelaide Local Health Network, Woodville, South Australia
  - Alfred Heath, Melbourne, Victoria
  - Eastern Clinical Research Unit, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] McAlpine FE, Lee JK, Harms AS, Ruhn KA, Blurton-Jones M, Hong J, Das P, Golde TE, LaFerla FM, Oddo S, Blesch A, Tansey MG. Inhibition of soluble TNF signaling in a mouse model of Alzheimer's disease prevents pre-plaque amyloid-associated neuropathology. Neurobiol Dis. 2009 Apr;34(1):163-77. doi: 10.1016/j.nbd.2009.01.006. PMID 19320056
- [Result] Cavanagh C, Tse YC, Nguyen HB, Krantic S, Breitner JC, Quirion R, Wong TP. Inhibiting tumor necrosis factor-alpha before amyloidosis prevents synaptic deficits in an Alzheimer's disease model. Neurobiol Aging. 2016 Nov;47:41-49. doi: 10.1016/j.neurobiolaging.2016.07.009. Epub 2016 Jul 25. PMID 27552480
- [Result] Sama DM, Mohmmad Abdul H, Furman JL, Artiushin IA, Szymkowski DE, Scheff SW, Norris CM. Inhibition of soluble tumor necrosis factor ameliorates synaptic alterations and Ca2+ dysregulation in aged rats. PLoS One. 2012;7(5):e38170. doi: 10.1371/journal.pone.0038170. Epub 2012 May 29. PMID 22666474
- [Result] MacPherson KP, Sompol P, Kannarkat GT, Chang J, Sniffen L, Wildner ME, Norris CM, Tansey MG. Peripheral administration of the soluble TNF inhibitor XPro1595 modifies brain immune cell profiles, decreases beta-amyloid plaque load, and rescues impaired long-term potentiation in 5xFAD mice. Neurobiol Dis. 2017 Jun;102:81-95. doi: 10.1016/j.nbd.2017.02.010. Epub 2017 Feb 24. PMID 28237313
- See also: Related Info — http://www.inmunebio.com
- See also: Part the cloud grant information - Alzheimer's Association — https://www.alz.org/partthecloud/research.asp